CLINICAL TRIAL: NCT04278157
Title: A Culturally Centered CBT Protocol for Suicidal Ideation and Suicide Attempts Among Latinx Youth
Brief Title: Culturally Centered CBT for Latinx Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bradley Hospital (Other)
Collaborators: Brown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1437564-1
Record Dates: First submitted 2020-02-13; First posted 2020-02-20 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Suicide
Keywords: Suicidal Ideation; Suicide Attempt; Latina, Latino, Latinx youth
MeSH Terms: conditions — Suicide; Suicidal Ideation; Suicide, Attempted | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SCBT-SB (Experimental): A culturally centered CBT treatment protocol called Socio-Cognitive Behavioral Therapy for Suicidal Behavior (SCBT-SB)
  Interventions: Behavioral: Socio-Cognitive Behavioral Therapy for Suicidal Behavior (SCBT-SB)
- Treatment as Usual (Active Comparator): Treatment as usual is base on the standard care for teens and their parents under a community mental health center.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Socio-Cognitive Behavioral Therapy for Suicidal Behavior (SCBT-SB) — The SCBT-SB is a manualized and flexible intervention that uses a modular approach to the treatment of adolescent suicidality. After the first mandatory module (Crisis module), and at the end of each subsequent module, the therapist works with the teen and caregivers to determine the next one. The Crisis Module is fixed and represent the intervention core skills with 9 sessions. The optional coping skills modules include Thoughts, Emotional Regulation, Family Communication, Social Interaction, Activity, Trauma, and Substance Use.
  Arms: SCBT-SB
Behavioral: Treatment as Usual — Therapy that typically consist of eclectic individual therapy including CBT, emphasizing psychoeducation and providing support, with occasional conjoint parent sessions or individual caregiver sessions. The treatment as usual primarily focuses on generating solutions to the adolescent and caregivers most urgent concerns.
  Arms: Treatment as Usual

SUMMARY:
The primary aim of the proposed research is to test the effect of a culturally centered treatment protocol, the Socio-cognitive behavioral therapy (SCBT), versus Treatment as Usual on suicidal thoughts and attempts, and depressive symptoms, in a clinical sample of Latinx adolescents. The study is trying to determine, if we take into account perspectives of Latin immigrant families and minority youth, whether better outcomes can be found for this high risk group.

DETAILED DESCRIPTION:
The overall goal of this research program is to provide effective culturally relevant care to Latin families, and address the National Institute on Minority Health and Health Disparities (NIMHD) mission of reducing disparities in underserved and minority populations. Evidence-based and culturally centered treatments for Latinx teens (Latinx = gender inclusive term) with suicidal ideation and attempts (SIA) and their families are quite limited. Emerging evidence indicate that Cognitive behavioral therapy (CBT) is a promising treatment approach in reducing suicidal ideation and attempts in Non-Latinx White adolescents. However, culturally adapted treatments have been shown to benefit Latin families more that non-culturally adapted treatments. This study is innovative in its use of a culturally centered CBT treatment protocol (Socio-Cognitive Behavioral Therapy for Suicidal Behavior-SCBT-SB) to address the specific needs of Latinx teens and their families. The SCBT-SB, is a modified version of two CBT protocols, which addresses central issues in adolescent identity formation (e.g. ethnicity, sexual orientation), family interactions and communication, and parenting skills. The SCBT-SB was developed with Latinx youth with SIA in Puerto Rico and further modified for Latin families in the US. Feasibility of this modified version of the SCBT-SB was tested in the US by conducting a pilot randomized clinical trial (RCT) (n=46) of SCBT vs treatment-as-usual (TAU) with positive results. It was found that SCBT-SB was feasible to implement in a community mental health center with frontline therapists, acceptable to families, and showed reductions in suicidal ideation and depressive symptoms. The scientific premise of the proposed study is that immigration and acculturation (the process of assimilation to the host culture) and enculturation (maintaining cultural values and costumes) experiences have an impact on SIA in Latinx teens; and that personalization of an evidence-based treatment, according to cultural and immigration experiences, will result in better treatment outcomes than TAU. This application proposes a hybrid efficacy/effectiveness trial with 160 suicidal Latinx teens randomly assigned, following baseline assessment, to 2 treatment conditions, TAU and SCBT-SB. Follow-up assessment will take place at 3, 6 and 12 months after baseline. All treatment will take place at a community mental health clinic. The specific aims are: 1) To test the effect of the SCBT-SB versus TAU on suicidal ideation in a clinical sample of adolescents under conditions of strong external validity, and 2) To test the effect of the SCBT-SB versus TAU on depressive symptoms, given its high correlation with SIA. Exploratory aims are: 3) To examine the effect of SCBT-SB versus TAU on suicide attempts, and 4) To examine potential mediators (family environment) of treatment outcome. Successful completion of this study will positively impact treatment of Latinx immigrant adolescents at high risk of SIA in the US.

ELIGIBILITY:
Inclusion Criteria:

* Latinx, defined as have been born in a Latin country or having at least one biological parent, grandparent or an ancestor that was born in a Latin country
* Severe Suicidal Ideation (SI), defined as a score of 22 or above on the SIQ-JR or having made a Suicide Attempts (SA) within the last 3 months
* Caregivers and adolescents fluent in Spanish or English language and legal guardian willing to participate

Exclusion Criteria:

* psychosis
* substance use disorder, rated severe on the DSM-5
* cognitive impairment represented by an IQ below 85

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 114 (Actual)
Dates: Start 2020-02-27 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
Suicidal ideation | Change from baseline to 3 month, 6 month, and 12 month follow up points.
  Suicidal ideation measured using the Suicide Ideation Questionnaire-Junior (SIQ-JR), the minimum score is 0 and the maximum 90. A higher score represents increase severity and frequency of suicidal thoughts.
Depressive symptoms by self-report | Change from baseline to 3 month, 6 month, and 12 month follow up points.
  Level of depressive symptomatology using the Children Depression Inventory 2 (CDI-2), the minimum score is 0 and the maximum 56. A higher score means higher level of depressive symptoms.
Depressive symptoms by clinical interview | Change from baseline to 3 month, 6 month, and 12 month follow up points.
  Depressive symptoms using the Children's Depression Rating Scale-Revised (CDRS-R), the minimum raw score is 17 and the maximum 113. A higher score means higher level of depressive symptoms.

SECONDARY OUTCOMES:
Suicide Attempts | Change from baseline to 6 months follow-up
  Number of total actual and interrupted suicide attempts using the Columbia-Suicide Severity Rating Scale (C-SSRS)
Suicide Attempts | Change from 6 months to 12 months follow-up
  Actual and interrupted suicide attempts (yes or no) using the Columbia-Suicide Severity Rating Scale (C-SSRS)
Suicide Attempts | Change from baseline to 12 months follow-up
  Actual and interrupted suicide attempts (yes or no) using the Columbia-Suicide Severity Rating Scale (C-SSRS)

CONTACTS AND LOCATIONS:
Overall Officials: Yovanska Duarte-Velez, PhD, Principal Investigator — Bradley Hospital
Locations (2):
- United States (2):
  - Hasbro Children's Hospital (Inpatient Psychiatric Unit), Providence, Rhode Island
  - Bradley Hospital, Riverside, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available to other researchers by request and as per NIH data sharing guidelines. The PI will also consult to anyone interested in replicating the intervention and study.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: One year following collection and final analyses.
Access Criteria: By email contact with PI.

REFERENCES:
- [Background] Duarte-Velez Y, Torres-Davila P, Spirito A, Polanco N, Bernal G. Development of a treatment protocol for Puerto Rican adolescents with suicidal behaviors. Psychotherapy (Chic). 2016 Mar;53(1):45-56. doi: 10.1037/pst0000044. PMID 26928136
- [Background] Duarte-Velez Y, Jimenez-Colon G, Jones RN, Spirito A. Socio-Cognitive Behavioral Therapy for Latinx Adolescent with Suicidal Behaviors: A Pilot Randomized Trial. Child Psychiatry Hum Dev. 2024 Jun;55(3):754-767. doi: 10.1007/s10578-022-01439-z. Epub 2022 Oct 1. PMID 36183051